CLINICAL TRIAL: NCT06500546
Title: The Effect of Different Adhesion Strategies on the Clinical Success of Non-caries Cervical Restorations.
Brief Title: The Effect of Different Adhesion Strategies on the Clinical Success
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Demirci, Prof.Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/58
Record Dates: First submitted 2024-06-28; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Poor Aesthetic of Existing Restoration of Tooth; Dental Restoration Failure of Marginal Integrity; Unacceptable Morphology of Tooth Restoration; Secondary Caries

STUDY DESIGN:
Intervention Model Description: comparison of restoration success
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesion Strategies (Other): Four non-carious cervical lesions from patients will be separated into four groups according to differnet adhesion strategies
  Interventions: Procedure: Treatment of cervical lesions
- Different procedure (Other): All lesions to which adhesives are applied according to different adhesion strategies will be restored with the same type of composite material.
  Interventions: Procedure: Treatment of cervical lesions

INTERVENTIONS:
Procedure: Treatment of cervical lesions — Four non-carious cervical lesions from patients will be separated into four groups according to according to the adhesion trategies described below:
  1. adhesive material will be applied in total-etch mode,
  2. adhesive material will be applied in self-etch,
  3. universal adhesive material will be applied for 10 sec. in total-etch mode, which includes rubbing,
  4. universal adhesive material will be applied for 10 sec. in self-etch mode, which includes rubbing,
  Other Names: differnet adhesion procedures

SUMMARY:
The study will involve 41 people who regularly seek treatment at clinics. Participants must be in generally good health and be older than eighteen. must have at least 20 teeth in an occlusion and maintain appropriate dental hygiene. They have to be treated for a minimum of four non-cancerous cervical lesions in their mouths.Four non-carious cervical lesions from patients will be separated into four groups, and adhesive material will be applied to the lesions in each group using different procedures. Evaluation will be performed based on World Dental Federation (FDI) criteria after initial, ½, 1, 2, 3, 4, and 5 years.

DETAILED DESCRIPTION:
The study will involve 41 people who regularly seek treatment at clinics. Participants must be in generally good health and be older than eighteen. must have at least 20 teeth in an occlusion and maintain appropriate dental hygiene. They have to be treated for a minimum of four non-cancerous cervical lesions in their mouths.Four non-carious cervical lesions from patients will be separated into four groups, and adhesive material will be applied to the lesions in each group using different procedures. Evaluation will be performed based on World Dental Federation (FDI) criteria after initial, ½, 1, 2, 3, 4, and 5 years. In each evaluation period, esthetic (surface gloss, surface coloration, marginal discoloration, color match and translucency, esthetic anatomic form), functional (fracture and retention, marginal adaptation), and biologic criteria (postoperative sensitivity and vitality, caries recurrence) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Good oral hygiene normal occlusal relationship with natural dentition
* At least 20 teeth are in occlusion The tooth with the lesion must be vital. non-mobile and non-carious
* Accepts Healthy Volunteers

Exclusion Criteria:

under the age of 18

* Poor oral hygiene poor general health condition
* Bruxism or uncontrolled parafunction
* Patients with periodontal or gingival diseases

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
retention rate of restorations | Restorations will be evaluated 1 week, 6 months, 12 months and 24 months after finishing.
  survival of restorations discoloration, color match, translucency, esthetic anatomic form), functional (fracture and retention, marginal adaptation), and biologic criteria (postoperative sensitivity). and vitality, caries recurrence)

SECONDARY OUTCOMES:
retention rate of restorations | Restorations will be evaluated 36 months, 48 months and 60 months after finishing.
  survival of restorations discoloration, color match, translucency, esthetic anatomic form), functional (fracture and retention, marginal adaptation), and biologic criteria (postoperative sensitivity). and vitality, caries recurrence)

IPD SHARING:
Plan to Share IPD: No